CLINICAL TRIAL: NCT05742295
Title: Preventing Cefoperazone/Sulbactam Induced Coagulopathy in Critically Ill Egyptian Patients: Efficacy of Vitamin K Prophylactic Doses
Brief Title: Prevention of Cefoperazone-induced Coagulopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Hebatallah Ali Abdeen, Clinical pharmacist, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Vit. K for SULBinCo
Record Dates: First submitted 2023-02-10; First posted 2023-02-23 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Antibiotic Side Effect
Keywords: Coagulopathy; Cefoperazone; Vitamin K; Cefoperazone/sulbactam
MeSH Terms: conditions — Hemostatic Disorders | interventions — Vitamin K

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): vitamin K is used as a prophylactic dose to prevent cefoperazone/sulbactam coagulopathy.
  Interventions: Drug: Vitamin K
- Control group (No Intervention)

INTERVENTIONS:
Drug: Vitamin K — Coadministration of vitamin K with the first dose of cefoperazone/sulbactam
  Arms: Intervention group

SUMMARY:
Evaluating the effect of prophylactic doses of vitamin K in preventing the adverse effect of cefoperazone/sulbactam induced coagulopathy in critically ill patients.

DETAILED DESCRIPTION:
One of the most challenging issues in the intensive care unit is treating multidrug-resistant (MDR) bacterial infections weighing benefit to risk ratio. MDR bacterial infection in ICU is a major public health problem and the main cause of mortality in ICUs in Egypt. A study published in the American Journal of Infection Control pointed out that the prevalence of MDR bacterial infections in the ICU was 54%.

Cefoperazone is a 3rd generation cephalosporin antibiotic covering many Gram-positive and Gram-negative bacteria, sulbactam is a beta-lactamase inhibitor which is used in combination with many antibiotics to overcome beta-lactamase producing bacteria, therefore the combination of cefoperazone/sulbactam has activity against MDR gram-negative bacteria. On the other hand, cefoperazone has been shown to have the adverse effects of inducing coagulopathy which is reported in many case reports and retrospective cohort studies. In most cases, coagulopathy events occur within a few days from the start of using cefoperazone/sulbactam, therefore the ICU staff was obliged to discontinue the antibiotic and choose another alternative leading to increasing the risk of resistant bacteria and treatment failure. Therefore, discontinuing the antibiotic due to its serious adverse events will lead to poor outcomes, more bacterial resistance, and more cost therapeutic plans for treating the infection and managing the severe adverse drug events which have been occurred such as bleeding. There are 2 mechanisms for cefoperazone-induced coagulopathy. The first the mechanism is related to N-methylthiotetrazole (NMTT), a side chain in cefoperazone molecule, which is responsible for the inhibition of a vitamin K-dependent carboxylation process leading to antagonizing blood clotting factors. The the second mechanism is antibiotics, in general, kill the normal flora in the gut which produce vitamin K. This cefoperazone/sulbactam-induced coagulopathy is not found in healthy volunteers or patients with adequate vitamin K activity, therefore, could consider cefoperazone/sulbactam-induced coagulopathy in critically ill patients, as related to nutritional status of these patients specifically with regard to vitamin K. This study aimed at studying the effect of co-administration of prophylactic doses of vitamin k during the administration of cefoperazone/sulbactam to keep the normal daily requirements of vitamin k, therefore preventing coagulopathy.

ELIGIBILITY:
Inclusion Criteria:

* ICU admitted patients on treatment or prophylactic doses of cefoperazone/sulbactam.

Exclusion Criteria:

* Patients' aged <18 years
* Pregnancy or breastfeeding women
* Active bleeding or bleeding disorder
* Patients having an abnormal baseline coagulation profile.
* Patients administer total parenteral nutrition with regular vitamin k supplements.
* Refusal to sign the written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with changes in INR level | During the duration of cefoperazone/sulbactam treatment up to 2 weeks
  comparing INR level between baseline INR (before starting the antibiotic) and during the treatment with the antibiotic

SECONDARY OUTCOMES:
Number of Participants with bleeding incidence | During the duration of cefoperazone/sulbactam treatment up to 2 weeks
  Internal bleeding as hematemesis or melena

CONTACTS AND LOCATIONS:
Locations (1):
- 6-October Hospital, Giza, Egypt

REFERENCES:
- [Background] Cai Z, Yang W, He Y, Chen Q, Wang S, Luo X, Wang X. Cefoperazone/Sulbactam-Induced Abdominal Wall Hematoma and Upper Gastrointestinal Bleeding: A Case Report and Review of the Literature. Drug Saf Case Rep. 2016 Dec;3(1):2. doi: 10.1007/s40800-016-0025-9. PMID 27747682
- [Background] Schentag JJ, Welage LS, Grasela TH, Adelman MH. Determinants of antibiotic-associated hypoprothrombinemia. Pharmacotherapy. 1987;7(3):80-6. doi: 10.1002/j.1875-9114.1987.tb03522.x. PMID 3306622
- [Background] Schentag JJ, Welage LS, Williams JS, Wilton JH, Adelman MH, Rigan D, Grasela TH. Kinetics and action of N-methylthiotetrazole in volunteers and patients. Population-based clinical comparisons of antibiotics with and without this moiety. Am J Surg. 1988 May 31;155(5A):40-4. doi: 10.1016/s0002-9610(88)80210-1. PMID 3163900
- [Background] Allison PM, Mummah-Schendel LL, Kindberg CG, Harms CS, Bang NU, Suttie JW. Effects of a vitamin K-deficient diet and antibiotics in normal human volunteers. J Lab Clin Med. 1987 Aug;110(2):180-8. PMID 3598347
- [Background] Mendes R, Policarpo S, Fortuna P, Alves M, Virella D, Heyland DK; Portuguese NUTRIC Study Group. Nutritional risk assessment and cultural validation of the modified NUTRIC score in critically ill patients-A multicenter prospective cohort study. J Crit Care. 2017 Feb;37:45-49. doi: 10.1016/j.jcrc.2016.08.001. Epub 2016 Aug 10. PMID 27621112
- [Background] Fouda R, Soliman MS, ElAnany MG, Abadeer M, Soliman G. Prevalence and risk factors of MRSA, ESBL and MDR bacterial colonization upon admission to an Egyptian medical ICU. J Infect Dev Ctries. 2016 Apr 28;10(4):329-36. doi: 10.3855/jidc.6798. PMID 27130993
- [Background] Abdelkader MM, Aboshanab KM, El-Ashry MA, Aboulwafa MM. Prevalence of MDR pathogens of bacterial meningitis in Egypt and new synergistic antibiotic combinations. PLoS One. 2017 Feb 16;12(2):e0171349. doi: 10.1371/journal.pone.0171349. eCollection 2017. PMID 28207768
- [Background] Talaat M, El-Shokry M, El-Kholy J, Ismail G, Kotb S, Hafez S, Attia E, Lessa FC. National surveillance of health care-associated infections in Egypt: Developing a sustainable program in a resource-limited country. Am J Infect Control. 2016 Nov 1;44(11):1296-1301. doi: 10.1016/j.ajic.2016.04.212. Epub 2016 Jun 20. PMID 27339791
- [Background] Hu HR. Fatal Vitamin K-Dependent Coagulopathy Associated with Cefoperazone/Sulbactam: A Case Report. Drug Saf Case Rep. 2019 Jun 14;6(1):6. doi: 10.1007/s40800-019-0100-0. PMID 31201572
- [Background] Wang W, Liu Y, Yu C, Tan J, Xiong W, Dong D, Li S, Zhang R, Li J, Wu Y, Zong Z, Su N, Zou K, Wu G, Sun X. Cefoperazone-sulbactam and risk of coagulation disorders or bleeding: a retrospective cohort study. Expert Opin Drug Saf. 2020 Mar;19(3):339-347. doi: 10.1080/14740338.2020.1713090. Epub 2020 Jan 27. PMID 31914329
- [Background] Park GH, Kim S, Kim MS, Yu YM, Kim GH, Lee JS, Lee E. The Association Between Cephalosporin and Hypoprothrombinemia: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2019 Oct 16;16(20):3937. doi: 10.3390/ijerph16203937. PMID 31623191